CLINICAL TRIAL: NCT07211139
Title: Head and Neck Advanced Research for Multi-Omics and Optimized Immunotherapy(HARMONI)
Brief Title: Head and Neck Advanced Research for Multi-Omics and Optimized Immunotherapy
Acronym: HARMONI
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JinYong Kim, Assistant Clinical Professor, Department of Oncology, Samsung Medical Center, Samsung Medical Center
Other Study IDs: 2025-04-059
Record Dates: First submitted 2025-09-17; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Biospecimen Description:
  Tumor tissue and peripheral blood samples will be collected for translational research.
  Tumor tissue: Paired biopsies will be obtained from lesions identified by medical oncologists and otolaryngologists. Sampling will occur before treatment, after one cycle (3 ± 1 weeks), and, if feasible, at disease progression. Fresh frozen tissue will be prioritized; if unavailable, formalin-fixed paraffin-embedded (FFPE) tissue will be used.
  Peripheral blood: 20-30 mL will be collected at baseline, 3, 6, and 12 weeks after treatment initiation, during radiologic assessments, and at disease progression. Each participant will have at least six blood draws.
  Stored sample types: Fresh frozen tumor tissue, FFPE tissue, whole blood, plasma, serum, and peripheral blood mononuclear cells (PBMCs).
  All biospecimens will be stored under controlled conditions for immunologic, genomic, and molecular analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head and neck squamous cell carcinoma is a heterogeneous cancer with varying prognoses depending on anatomical location and characteristics, and advanced cancers have a poor prognosis. This study aimed to examine changes in the tumor microenvironment and systemic immune system before and after combination therapy with immune checkpoint inhibitors, the standard first-line treatment for head and neck cancer. The rationale for this research and development project is as follows:

1. While immune checkpoint inhibitors have improved survival rates for head and neck cancer patients, they are only effective in approximately 15% of patients. Because biomarkers predicting treatment response have not yet been clearly identified, targeting target patient populations is challenging.
2. While numerous studies have examined the tumor microenvironment in head and neck cancer, no studies have spatially compared dynamic changes before and after immune checkpoint inhibitor treatment using paired tissue and blood biopsies. Therefore, the specific treatment mechanisms remain unclear.
3. Little is known about how changes in the tumor microenvironment are reflected in the peripheral blood, making noninvasive treatment response monitoring difficult.
4. Immune checkpoint inhibitor treatment is known to enhance the efficacy of subsequent taxane-based chemotherapy, but the mechanism remains unknown.

Therefore, we aim to explore biomarkers that predict treatment response to combination therapy with immune checkpoint inhibitors and cytotoxic chemotherapy in patients with advanced/metastatic head and neck cancer and develop personalized treatment strategies.

DETAILED DESCRIPTION:
1. Background 1.1 Research Background Immune checkpoint inhibitors (ICIs) have emerged as a new class of anticancer therapy following cytotoxic chemotherapy and targeted therapy. They have demonstrated survival benefits in various solid tumors, including head and neck cancers, thereby shifting the paradigm of cancer treatment. Tumors evade immune surveillance through checkpoint molecules such as PD-1 and CTLA-4, and the development of ICIs such as pembrolizumab and nivolumab has shown efficacy in head and neck cancers as well.

Advanced and metastatic head and neck cancers not only pose life-threatening risks but also severely affect speech, swallowing, and appearance, leading to a higher suicide rate compared to the general population. In Korea, the incidence of head and neck cancer increased by about 30% between 2010 and 2020, with tongue cancer showing a particularly steep rise of 7.7% per year in young adults aged 20-30.

In the KEYNOTE-048 trial, pembrolizumab combined with platinum-based chemotherapy significantly prolonged overall survival compared to cetuximab-based regimens, with greater benefit observed in patients with PD-L1 CPS ≥20 or ≥1. Subsequent analyses showed that the survival benefit correlated with PD-L1 CPS only in the pembrolizumab-combination group, and about 20% of patients were identified as long responders. However, the overall response rate to ICIs remains only 15-26%, and PD-L1 CPS alone does not fully explain treatment outcomes.

The TIME (tumor immune microenvironment) study on head and neck cancer classified tumors into fully infiltrated, stroma-restricted, immune-excluded, and immune-desert subtypes, with 48% being fully infiltrated. Tumors with high expression of cytokines such as CXCL13, IFN-γ, and IL-10 exhibited more active immune cell infiltration. However, these results were based on pre-treatment tissues, and there is a lack of studies investigating TIME changes after treatment.

In recurrent head and neck cancer, intratumoral and stromal TIL density significantly decreased, while the proportion of immune-desert tumors increased. Stromal TIL enrichment correlated with better response to ICIs. However, this study was based on AI-driven image analysis and did not capture detailed immune microenvironment composition or post-treatment dynamics.

In Japan, spatial transcriptomics analysis was performed in one head and neck cancer patient treated with nivolumab, revealing that post-treatment loss of MHC class I gene expression was associated with immune resistance.

High CXCL13 expression is linked to the formation of tertiary lymphoid structures (TLS) and strongly associated with immune cell distribution in the TIME. TCGA analyses showed that CXCL13 expression is significantly higher in head and neck cancers compared to normal tissues, and correlates with the abundance of CD8+ T cells, B cells, macrophages, and other immune cells. Thus, it is necessary to investigate whether CXCL13 and TLS change following ICI treatment. In addition, CD44+ cancer stem cells in head and neck cancer are associated with poor prognosis, and their dynamic changes before and after immunotherapy warrant investigation.

Peripheral blood-based approaches to predict immune responses have also been explored. Retrospective studies using inflammatory markers such as NLR, MLR, and PLR developed predictive models that outperformed PD-L1 CPS in accuracy. Another study reported that PD-L1 expression on monocytes after chemoradiotherapy correlated with plasma CXCL11 levels. Gene expression analyses of pre- and post-surgical samples identified significant differences in EIF2, EIF4, and mTOR signaling pathways. Moreover, cytokine levels in the serum of head and neck cancer patients were significantly higher than in healthy controls, and an increase in immature neutrophils was suggested to be associated with tumor infiltration.

In a follow-up analysis of the KEYNOTE-048 trial, patients treated with pembrolizumab plus chemotherapy exhibited longer progression-free survival with subsequent taxane therapy (PFS2), independent of PD-L1 CPS (HR 0.67, P=0.00788). This suggests that ICI treatment may enhance responsiveness to later taxane-based chemotherapy. Biomarker studies are needed to explain these interactions, and given regional and ethnic variations, research based on Korean patients is particularly important.

1.2 Research Summary Head and neck squamous cell carcinoma (HNSCC) is a heterogeneous malignancy with prognosis varying by anatomical site and tumor characteristics, but advanced disease generally carries poor outcomes. This study aims to investigate dynamic changes in both the tumor immune microenvironment (TIME) and systemic immunity before and after first-line ICI plus chemotherapy in HNSCC patients.

The rationale for this project is as follows:

1. ICIs have improved survival in HNSCC but remain effective in only about 15% of patients. Predictive biomarkers to select responders remain unclear.
2. Although many studies have investigated TIME in HNSCC, no study has performed paired analyses of tumor tissue and blood before and after ICI treatment to assess spatial and temporal immune changes.
3. The extent to which TIME changes are reflected in peripheral blood remains unknown, limiting non-invasive monitoring of treatment response.
4. ICIs are known to enhance the efficacy of subsequent taxane chemotherapy, but the underlying mechanism is not understood.

Therefore, this study seeks to identify predictive biomarkers for treatment response and develop personalized therapeutic strategies for patients with advanced or metastatic HNSCC receiving ICI plus chemotherapy.

* Study Objectives and Goals To identify predictive biomarkers of treatment response and develop personalized therapeutic strategies in patients with advanced/metastatic HNSCC treated with ICIs plus chemotherapy.

  ________________________________________
* Study Duration The study will be conducted for 3 years from the date of IRB approval. Participants will be followed for 3 years from enrollment. Analyses will begin in the second year, focusing on dynamic changes in the TIME and systemic immunity before and after treatment. In the third year, biomarkers of ICI response and resistance will be identified, and correlations between TIME and systemic immune changes will be evaluated.

  ________________________________________
* Study Participants 4.1 Inclusion and Sample Size Justification The study aims to explore immune microenvironment (TME) changes observed in tumor samples before and after ICI-based treatment. The primary outcome is to assess changes in immune cell marker expression and their association with treatment response. This exploratory design seeks to generate clinically meaningful immunologic patterns as preliminary data for future studies (e.g., biomarker-driven predictive model development, prospective validation).

Eligible patients will be those diagnosed with advanced/metastatic HNSCC receiving first-line ICI plus chemotherapy. Approximately 30 paired pre- and post-treatment samples will be collected.

The target sample size of 30 patients is based on feasibility considerations (availability of paired samples, recruitment within 1.5-2 years) and aligns with prior studies of similar design, which typically included 20-40 patients. This is deemed an appropriate exploratory cohort size for the study objectives.

At Samsung Medical Center, about 600 HNSCC patients are treated annually, with over 50 newly diagnosed advanced/metastatic cases receiving palliative chemotherapy each year, ensuring sufficient patient accrual for this study.

5 Study Design and Methods 5.1 Dynamic Analysis of Immune Changes Before and After Treatment

* Tumor Immune Microenvironment (TIME) Analysis Paired tumor biopsies or FFPE samples will be collected before and after treatment, sectioned, and analyzed. Immune biomarkers to be evaluated include tumor cells, T cells, B cells, neutrophils, macrophages, immune gene signatures (e.g., interferons such as IFN-γ, and interleukin families), T-cell subsets (CD4+, CD7+, CD8+, CD16, CD34+, CD38+, CD56+), cancer stem cells (CD44), CXCL13, and PD-1/PD-L1 expression. Changes in these biomarkers will be compared pre- and post-treatment. Interactions between tumor and immune cells will be examined, as well as alterations in specific immune cell clusters and spatial patterns (e.g., tertiary lymphoid structures, immune hubs). Additionally, extracellular vesicle changes will be evaluated to explore mechanisms underlying enhanced responsiveness to subsequent taxane therapy after ICI treatment.
* Systemic Immunity Analysis Peripheral blood mononuclear cells (PBMCs) will be isolated from blood samples and analyzed using flow cytometry. Existing validated panels in the PI's laboratory will be adapted for this study. Quantitative changes in immune cell populations and cytokines (e.g., IFN-γ) before and after treatment will be assessed.

5.2 Development of a Personalized Treatment Strategy for ICIs in Head and Neck Cancer

* Identification of Predictive Biomarkers Clinical response data to ICI therapy will be integrated with tissue and blood-based analyses to identify candidate predictive biomarkers. Significant immune cell changes will be defined as ≥1.5-fold differences. Predictive models will be developed using multivariate and regression analyses, with the goal of achieving an Area Under the Curve (AUC) ≥0.80.
* Correlation Between TIME and Systemic Immunity Associations between tumor microenvironmental changes and peripheral blood changes will be examined. A Pearson correlation coefficient ≥0.5 will be considered meaningful. Further, the relationship between these immunologic changes and patient prognosis will be evaluated.
* Mechanisms of ICI Resistance Comparative analyses between responders and non-responders will be conducted to elucidate mechanisms of primary resistance. When feasible, paired tumor and blood samples at the time of disease progression will also be analyzed to investigate mechanisms of acquired resistance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent/metastatic head and neck squamous cell carcinoma (HNSCC)
* Received first-line combination therapy with immune checkpoint inhibitor and cytotoxic chemotherapy
* Availability of tumor tissue samples at Samsung Medical Center
* p16 and PD-L1 expression status evaluable within the institution
* Age ≥ 20 years
* Ability to understand the study purpose and provide written informed consent

Exclusion Criteria:

* Not meeting the inclusion criteria
* Considered ineligible for enrollment at the discretion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent or metastatic head and neck squamous cell carcinoma treated at Samsung Medical Center. Approximately 600 patients with head and neck cancer visit the center annually, and more than 50 patients are newly diagnosed with recurrent/metastatic disease and receive systemic therapy each year. This study will recruit eligible patients from this population.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 3 years after enrollment.
  Time from initiation of treatment to death from any cause. Estimated using Kaplan-Meier survival analysis. The effect of clinical and treatment variables on survival will be evaluated using the Cox proportional hazards model.
Treatment Response | From treatment initiation until disease progression or death, whichever occurs first, assessed every 6-12 weeks, up to 36 months.
  Tumor response evaluated according to RECIST v1.1 criteria (Complete Response, Partial Response, Stable Disease, Progressive Disease).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Time Frame: Up to 3 years after enrollment.
  Time from initiation of treatment to disease progression or death. Kaplan-Meier method and Cox proportional hazards model.
Treatment Toxicity | From first dose of study treatment until 90 days after the last dose of study treatment, up to 36 months.
  Adverse events will be assessed and graded according to CTCAE criteria.
Between Clinical/Immunologic Variables and Treatment Outcomes | Up to 3 years after enrollment.
  Continuous variables will be compared using independent-sample t-test or Wilcoxon rank-sum test; categorical variables will be compared using chi-square test or Fisher's exact test. p-values <0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Privacy and Security IPD information represents and individual's characteristics, so sharing it mayy pose a risk of personal information leakage.

REFERENCES:
- [Background] Braakhuis BJ, Graveland AP, Dijk F, Ylstra B, van Wieringen WN, Leemans CR, Brakenhoff RH. Expression signature in peripheral blood cells for molecular diagnosis of head and neck squamous cell carcinoma. Oral Dis. 2013 Jul;19(5):452-5. doi: 10.1111/odi.12019. Epub 2012 Oct 3. PMID 23034102
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] Fang R, Chen Y, Huang B, Wang Z, Zhu X, Liu D, Sun W, Chen L, Zhang M, Lyu K, Lei W. Predicting response to PD-1 inhibitors in head and neck squamous cell carcinomas using peripheral blood inflammatory markers. Transl Oncol. 2025 Jan;51:102222. doi: 10.1016/j.tranon.2024.102222. Epub 2024 Dec 1. PMID 39616985
- [Background] Harrington KJ, Burtness B, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Brana I, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Lin J, Gumuscu B, Swaby RF, Rischin D. Pembrolizumab With or Without Chemotherapy in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma: Updated Results of the Phase III KEYNOTE-048 Study. J Clin Oncol. 2023 Feb 1;41(4):790-802. doi: 10.1200/JCO.21.02508. Epub 2022 Oct 11. PMID 36219809
- [Background] Idel C, Fleckner J, Plotze-Martin K, Werner L, Rades D, Theodoraki MN, Hofmann L, Huber D, Leichtle A, Hoffmann TK, Bruchhage KL, Pries R. Partial recovery of peripheral blood monocyte subsets in head and neck squamous cell carcinoma patients upon radio(chemo)therapy is associated with decreased plasma CXCL11. BMC Cancer. 2024 Apr 12;24(1):459. doi: 10.1186/s12885-024-12177-x. PMID 38609887
- [Background] Ishida Y, Agata Y, Shibahara K, Honjo T. Induced expression of PD-1, a novel member of the immunoglobulin gene superfamily, upon programmed cell death. EMBO J. 1992 Nov;11(11):3887-95. doi: 10.1002/j.1460-2075.1992.tb05481.x. PMID 1396582
- [Background] Iwasa YI, Nakajima T, Hori K, Yokota Y, Kitoh R, Uehara T, Takumi Y. A Spatial Transcriptome Reveals Changes in Tumor and Tumor Microenvironment in Oral Cancer with Acquired Resistance to Immunotherapy. Biomolecules. 2023 Nov 22;13(12):1685. doi: 10.3390/biom13121685. PMID 38136558
- [Background] Jung YS, Lee D, Jung KW, Cho H. Long-term Survivorship and Non-cancer Competing Mortality in Head and Neck Cancer: A Nationwide Population-Based Study in South Korea. Cancer Res Treat. 2023 Jan;55(1):50-60. doi: 10.4143/crt.2021.1086. Epub 2022 Mar 4. PMID 35698446
- [Background] Jung YS, Seok J, Hong S, Ryu CH, Ryu J, Jung KW. The emergence of oral cavity cancer and the stabilization of oropharyngeal cancer: Recent contrasting epidemics in the South Korean population. Cancer. 2021 May 15;127(10):1638-1647. doi: 10.1002/cncr.33434. Epub 2021 Feb 17. PMID 33595858
- [Background] Kim DH, Kang M, Park G, Mostafavi M, Lim Y, Ock CY, Koh J, Jeon YK, Jung KC, Ahn SH, Chung EJ, Kwon SK, Keam B. Changes in the tumor microenvironment in recurrent head and neck squamous cell carcinoma and its implication on efficacy of immune checkpoint inhibitors. Discov Oncol. 2024 Nov 20;15(1):686. doi: 10.1007/s12672-024-01504-0. PMID 39567471
- [Background] Leach DR, Krummel MF, Allison JP. Enhancement of antitumor immunity by CTLA-4 blockade. Science. 1996 Mar 22;271(5256):1734-6. doi: 10.1126/science.271.5256.1734. PMID 8596936
- [Background] Lin X, Zhao X, Chen Y, Yang R, Dai Z, Li W, Lin C, Cao W. CXC ligand 13 orchestrates an immunoactive microenvironment and enhances immunotherapy response in head and neck squamous cell carcinoma. Int J Immunopathol Pharmacol. 2024 Jan-Dec;38:3946320241227312. doi: 10.1177/03946320241227312. PMID 38252495
- [Background] Muijlwijk T, Nijenhuis DNLM, Ganzevles SH, Ekhlas F, Ballesteros-Merino C, Peferoen LAN, Bloemena E, Fox BA, Poell JB, Leemans CR, Brakenhoff RH, van de Ven R. Immune cell topography of head and neck cancer. J Immunother Cancer. 2024 Jul 24;12(7):e009550. doi: 10.1136/jitc-2024-009550. PMID 39053947
- [Background] Ouyang M, Sun H, Liu X, Wu H, Deng F, Shen E, Peng G, Wu H, Zhao Y, Xiong H, Liu B, He S, Hu Y, Liu P. The efficacy and safety of a taxane-based chemotherapy regimen combined with a PD-1 inhibitor in HNSCC: a multicenter real-world study. World J Surg Oncol. 2025 Jan 4;23(1):6. doi: 10.1186/s12957-024-03644-7. PMID 39754263
- [Background] Trellakis S, Farjah H, Bruderek K, Dumitru CA, Hoffmann TK, Lang S, Brandau S. Peripheral blood neutrophil granulocytes from patients with head and neck squamous cell carcinoma functionally differ from their counterparts in healthy donors. Int J Immunopathol Pharmacol. 2011 Jul-Sep;24(3):683-93. doi: 10.1177/039463201102400314. PMID 21978700
- [Background] Yu Y, Zakeri K, Sherman EJ, Lee NY. Association of Low and Intermediate Combined Positive Scores With Outcomes of Treatment With Pembrolizumab in Patients With Recurrent and Metastatic Head and Neck Squamous Cell Carcinoma: Secondary Analysis of Keynote 048. JAMA Oncol. 2022 Aug 1;8(8):1216-1218. doi: 10.1001/jamaoncol.2022.1846. PMID 35679031